CLINICAL TRIAL: NCT03159481
Title: Enhancing Glaucoma Medication Adherence Among African Americans
Brief Title: Glaucoma Management Optimism for African Americans Living With Glaucoma
Acronym: GOAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Laura E. Dreer, PhD, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9070592
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Usual Care + Health Promotion Intervention (Experimental): Usual glaucoma care along with telehealth-based brief culturally informed health promotion intervention
  Interventions: Behavioral: Usual Care + Health Promotion Intervention
- Usual Care Only (No Intervention): Usual glaucoma management only, no intervention.

INTERVENTIONS:
Behavioral: Usual Care + Health Promotion Intervention — Telephone sessions for approximately 5-6 weeks to enhance empowerment and skills for managing medication adherence.
  Other Names: GOAL
  Arms: Usual Care + Health Promotion Intervention

SUMMARY:
African Americans (AA) are at higher risk to develop and go blind from glaucoma than Caucasians. While glaucoma medications can help delay disease progression and possible blindness, problems with poor adherence have been documented for both racial groups, with a greater prevalence among AA. Of the very few interventions targeting glaucoma medication adherence studied to date, several methodological limitations persist. For example, few have been subjected to rigorous randomized clinical trial (RCT) designs, the intervention itself was designed and studied predominantly among Caucasians and thereby limiting generalizability, the effects on adherence have been short-term, most have been evaluated on small sample sizes, and/or the focus of the intervention was solely on providing patient education regarding eye disease and management. Needed in this important yet understudied area are culturally-relevant, health promotion-based approaches which are 1) targeted to high risk populations, 2) theoretically driven, 3) relevant to the beliefs, language, and values of underserved populations as well as challenges related to glaucoma medication adherence, 4) designed to promote preparation and readiness to engage in healthy behaviors, and 5) train patients in skills to use in order to more effectively problem-solve ongoing obstacles related to adherence.

The investigators published a paper in the Journal of Glaucoma investigating determinants related to objective medication adherence as measured by an electronic dosing aid (DA). Findings revealed poorer rates of adherence among AA patients with glaucoma compared to Caucasian patients with glaucoma. Evidence for racial differences in adherence have also been increasingly documented in the glaucoma literature. In a follow-up study with focus groups of AA's with glaucoma that was published in Optometry and Vision Sciences, the goal was to identify the specific barriers and facilitators related to glaucoma medication adherence among this high-risk group. Several key themes emerged such as patient, provider, and socioeconomic factors, along with barriers in views of health, perceived harm from treatment, costs, avoidant coping styles, forgetfulness, and in eyedrop administration/scheduling. The investigators used these results along with guidance from a consumer advisory board consisting of AA patients with glaucoma in order to develop and pilot test the resulting culturally relevant, health promotion-based intervention. The pilot data demonstrated feasibility and favorable preliminary efficacy for the intervention to significantly improve medication adherence to further pursue in a clinical trial.

DETAILED DESCRIPTION:
Aim 1: To evaluate the efficacy of a culturally relevant, health promotion-based intervention to increase rates of glaucoma medication adherence among AA patients with glaucoma as compared to usual care.

Aim 2: To longitudinally examine the associations between medical, demographic, cultural, socioeconomic, and ocular factors and objective medication adherence rates among AA's with glaucoma in the usual care only group. This aim will explore what factors are associated with glaucoma medication adherence, as defined by objective adherence measures, during usual care. This information will facilitate hypothesis generation and testing for future studies.

Aim 3: To longitudinally examine the associations between medical, demographic, cultural, socioeconomic, and ocular factors and objective medication adherence rates among AA's with glaucoma in the treatment arm (those receiving the treatment intervention). This aim will explore what patient-related factors are more or less likely to relate to the effectiveness of the intervention as defined by objective adherence. This information is useful for understanding which patients may ultimately most responsive to the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 21 years old
2. AA
3. have one of the following diagnoses: open-angle glaucoma, angle-closure glaucoma, glaucoma suspect, or ocular hypertension (OHTN) in one or both eyes
4. using or prescribed a topical prostaglandin analog
5. not to have undergone past laser or surgical glaucoma therapy within 3 months before the study
6. have two reliable visual fields over the past 2 years
7. English-speaking
8. cognitively oriented as defined by the Six-Item Screener (SIS) score of > 4 of 6
9. have access to a telephone,
10. agrees to random assignment to either arm of study
11. agrees to return for all follow-up visits
12. patient has been determined to be 80% or less adherent.

Exclusion Criteria:

1. cognitively unable to understand the study
2. does not instill their own eye drops
3. incapable of using the electronic MEMS bottle/cap after a brief practice session
4. known contraindications to Travoprost
5. has a severe hearing impairment impeding communication.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in medication rate adherence via an electronic dosing aid | Baseline, 3, 7 months, and 1 year
  Assessment in medication adherence will be obtained via an electronic dosing aid which tracks medication behavior (e.g., attempts to dispense eye drops).

SECONDARY OUTCOMES:
Knowledge of glaucoma management | Baseline, 3, 7 months, and 1 year
  This is an 11-item self-report measure of Patient Satisfaction with Glaucoma Treatment (Glaustat) that will be used to understand patients' knowledge of glaucoma and its management.
Glaucoma symptoms | Baseline, 3, 7 months, and 1 year
  The investigators will use the Glaucoma Symptom Scale to assess visual and nonvisual symptoms which developed from a modified version of a checklist used in the Ocular Hypertension Treatment Study. It has 10 items that ask respondents whether they have experienced certain symptoms (e.g., dryness) in the prior 4 weeks and to what extent they were bothered by these symptoms.
Health beliefs and illness perception | Baseline, 3, 7 months, and 1 year
  The 18-item Beliefs about Medicines Questionnaire (BMQ) will be used to assess patients' concerns about present/potential future adverse effects from their medications and their beliefs regarding the necessity of their medications. Scores are summed within each scale to create an overall scale score (range: 8-40 for a 'necessity scale' and 10-50 for a 'concerns scale'.
Social problem-solving skills | Baseline, 3, 7 months, and 1 year
  The Social Problem-Solving Inventory-Revised is a 25-item, self-report measure of motivation for solving problems and problem-solving abilities. The SPSI-R is based on a five dimensional model of problem-solving ability which includes two theoretically defined components, both of which will be measured: problem orientation and problem-solving skills.
Depressive symptomatology | Baseline, 3, 7 months, and 1 year
  The investigators will use the nine items of the Patient Health Questionnaire-9 (PHQ-9) scale to assess depressive symptomatology. The total score is calculated by summing each of the PHQ-9 items with higher scores indicating the presence of greater depressive symptomatology. The criterion, construct and external validity of the PHQ-9 have been well established using large medical samples.

OTHER OUTCOMES:
Sociodemographic variables | Baseline, 3, 7 months, and 1 year
  The investigators will evaluate the influence of several sociodemographic factors on outcomes (e.g., gender, income).
Medical factors | Baseline, 3, 7 months, and 1 year
  The investigators will also characterize ocular variables and other health related factors (e.g., intraocular pressure, degree of field loss, other medical conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dreer, Ph.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided